CLINICAL TRIAL: NCT03438162
Title: Impact of Pharmacotherapeutic Education on Medication Adherence and Adverse Outcomes in Type 2 Diabetes Mellitus Patients: Prospective, Randomized Study
Brief Title: Impact of Pharmacotherapeutic Education on Medication Adherence and Adverse Outcomes in Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Dubrava (Other)
Responsible Party: Principal Investigator, Srećko Marušić, Principal investigator, University Hospital Dubrava
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EDUDIABETES2017
Record Dates: First submitted 2017-09-20; First posted 2018-02-19 (Actual); Last update posted 2018-11-09 (Actual); Status verified 2018-11

CONDITIONS: Diabetes Mellitus, Type 2; Education; Drug-Related Side Effects and Adverse Reactions
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Drug-Related Side Effects and Adverse Reactions | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Patients in both groups received diabetes education during the hospital stay. Standardized diabetes education includes education regarding the disease, diet, physical activity, alcohol intake, smoking, education regarding diabetes medication, self monitoring of glucose, and education regarding acute and chronic complications.
- Intervention group (Experimental): Patients in both groups received diabetes education during the hospital stay. Standardized diabetes education includes education regarding the disease, diet, physical activity, alcohol intake, smoking, education regarding diabetes medication, self monitoring of glucose, and education regarding acute and chronic complications. Patients randomized in the intervention group received pre-discharge pharmacotherapeutic education. The education was conducted by a qualified physician.
  Interventions: Behavioral: Education

INTERVENTIONS:
Behavioral: Education — Patients randomized in the intervention group received pre-discharge pharmacotherapeutic education. The education was conducted by a qualified physician.
  Arms: Intervention group

SUMMARY:
Type 2 diabetes mellitus (T2DM) is a chronic progressive disease that affects more than 400 million people worldwide. There are a few studies evaluating ADRs in diabetics. Many patients experience ADRs soon after hospital discharge which can be attributed to the changes in the pharmacotherapy during hospitalization. Education and counseling of diabetic patients has been shown to improve medication adherence and clinical outcomes. Studies that included medical patients revealed that education can significantly reduce risk of ADRs after hospital discharge. Pharmacotherapeutic education is a part of comprehensive education of diabetics that is focused on a proper use of medications, prevention and early detection of ADRs.

DETAILED DESCRIPTION:
Type 2 diabetes mellitus (T2DM) is a chronic progressive disease that affects more than 400 million people worldwide. Besides adapting their lifestyle, a large majority of diabetic patients needs pharmacotherapy to achieve adequate glycaemic control. Additional pharmacotherapy is usually needed for the treatment of concomitant diseases and risk factors. This can result in polytherapy which puts patients et risk of adverse drug reactions (ADRs). There are a few studies evaluating ADRs in diabetics. A prospective observation study reported ADRs in 11.8% of diabetic patients in tertiary care hospital. Many patients experience ADRs soon after hospital discharge which can be attributed to the changes in the pharmacotherapy during hospitalization. These ADRs can result in early readmission and emergency department (ED) visits. In an Italian study, ADRs were reported in 73.8% of patients taking oral antidiabetics drugs within one month of study enrollment. It is estimated that between 11-38% of ambulatory ADRs are preventable. Medication adherence plays an important role in the treatment of T2DM because it clearly improves glycaemic control and clinical outcomes and lowers medical costs. Adherence rates to DM medications vary from 31% to 87% in retrospective studies and 53% to 98% in prospective studies. It is affected by many factors such as age, race, health beliefs, medication cost, co-pays, etc. Adherence is lower in the case of ADRs, when medications are taken more than twice daily, with concomitant depression and skepticism about the importance of medication. In recent years, 30-day readmission rate has been emphasised as a measure of healthcare quality. Diabetic patients have higher readmission rate compared to patients without DM. In the study by Ostling and al., 30-day readmission rate for patients with DM was 26%. Many readmissions are drug-related and can be caused by ADRs and non-adherence. These readmissions are potentially preventable. It is estimated that between 40%-57.1% of readmissions caused by ADRs and all readmissions caused by non-adherence are preventable. Education and counseling of diabetic patients has been shown to improve medication adherence and clinical outcomes. Studies that included medical patients revealed that education can significantly reduce risk of ADRs after hospital discharge. Pharmacotherapeutic education is a part of comprehensive education of diabetics that is focused on a proper use of medications, prevention and early detection of ADRs. The aim of this study was to evaluate the impact of pharmacotherapeutic education on 30-day post discharge medication adherence and adverse outcomes (ADRs, readmissions, ED visits and death) in diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older,
* diagnosis of T2DM and
* hospital discharge to the community.

Exclusion Criteria:

* cognitive disorders that would interfere with patient's participation,
* diagnosis of a terminal illness with a life expectancy <1 month,
* discharge to a long-term care facility or
* inability to be followed-up.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Medication adherence assessment method | one month
  The medication adherence of the two diabetic patients groups (intervention group and group without intervention) 30 days after the recruitment in the study was assessed by the pill count method. Where adherence was in the range from 80% to 100% the patients were categorized as adherent, and where adherence was less than 80% or more than 100% the patients were categorized as non-adherent.

SECONDARY OUTCOMES:
Adverse events questionnaire | one month
  The number of participants with treatment-related adverse events in the two diabetic patients groups (intervention group and group without intervention) 30 days after the recruitment in the study was compared using the questionnaire method which was conducted by the physician. The physician noted cause of the adverse event and marked its probability using the Naranjo adverse drug reaction probability scale. The Naranjo adverse drug reaction probability scale consists of 10 questions that are answered as either "Yes", "No", or "Do not know". Different point values (-1, 0, +1 or +2) are assigned to each answer. The adverse drug reaction is considered "definite" if the score is 9 or higher, "probable" if 5 to 8, "possible" if 1 to 4, and "doubtful" if 0 or less.

CONTACTS AND LOCATIONS:
Overall Officials: Srećko Marušić, Study Chair — University Hospital Dubrava
Locations (1):
- University Hospital Dubrava, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Marusic S, Melis P, Lucijanic M, Grgurevic I, Turcic P, Neto PRO, Bilic-Curcic I. Impact of pharmacotherapeutic education on medication adherence and adverse outcomes in patients with type 2 diabetes mellitus: a prospective, randomized study. Croat Med J. 2018 Dec 31;59(6):290-297. doi: 10.3325/cmj.2018.59.290. PMID 30610771